CLINICAL TRIAL: NCT06667518
Title: Reliability and Feasibility of Knee Traction Dynamometry and Electromyography Assessment in Children With Cerebral Palsy
Brief Title: Knee Neuromuscular Assessment in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, George Paras, Assistant Professor, University of Thessaly
Other Study IDs: neuromusc_knee_cp_child
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Force Measurement; Electromyography; Children; Cerebral Palsy; Lower Limb
Keywords: dynamometry; electromyography; cerebral palsy; child; lower limb
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Cerebral Palsy: Children with cerebral palsy, aged 5 to 16 years, classified at GMFCS levels I to III.
  Interventions: Device: Neuromuscular Activity Assessment

INTERVENTIONS:
Device: Neuromuscular Activity Assessment — K-Pull dynamometer is an assessment tool used to quantify muscle strength. It uses traction through a non-elastic strap to facilitate isometric contractions.
  K-Myo (non-invasive EMG sensor) is an assessment tool used to detect muscle activation and tracking patient's improvement.

SUMMARY:
The purpose of this study is to evaluate the reliability (intra-rater and inter-rater) of the K-Pull dynamometer and the K-Myo non-invasive electromyography sensor (assessing neuromuscular activity) in the evaluation of the lower limbs in children with cerebral palsy.

Specific objectives include:

* Examining differences in neuromuscular activity among children with CP classified at functional levels I to III on the GMFCS scale.
* Deriving conclusions from the correlation between electromyographic activity, muscle tone, and generated muscle strength.
* Assessing the applicability of neuromuscular activity assessment devices in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* children with spastic type cerebral palsy (CP),
* aged between 5 and 16 years,
* classified at GMFCS levels I to III,
* voluntary motor control,
* ambulatory, with or without the use of mobility aids,
* can understand and execute verbal commands.

Exclusion Criteria:

* have previously undergone interventions that affect neuromuscular performance (such as surgery or botulinum toxin injections)
* have sustained an injury,
* demonstrate a low level of compliance.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy, aged 5 to 16 years, classified at GMFCS levels I to III based on specific inclusion and exclusion criteria to ensure the reliability and feasibility of traction dynamometry and surface electromyography assessment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Through study completion, an average of 5 months
  Average Peak Force refers to the average highest force output recorded during isometric contractions and represents the maximal strength generated by the muscle group being assessed (e.g., hip or knee flexors and extensors). Unit of Measure: Newton (N)
Average Muscle Activation | Through study completion, an average of 5 months
  Average activation in the context of surface electromyography refers to the mean level of electrical activity detected from muscle fibers over a specific period. Unit of Measure: millivolt (mV)

SECONDARY OUTCOMES:
Muscle Tone | Through study completion, an average of 5 months
  Evaluated using the Modified Ashworth Scale. Unit of Measure: Scoring Options (0-4) // (higher scores - worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy - University of Thessaly, Lamia, Phthiotis, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulder-Brouwer AN, Rameckers EA, Bastiaenen CH. Lower Extremity Handheld Dynamometry Strength Measurement in Children With Cerebral Palsy. Pediatr Phys Ther. 2016 Summer;28(2):136-53. doi: 10.1097/PEP.0000000000000228. PMID 26744991
- [Background] Aertssen W, Smulders E, Smits-Engelsman B, Rameckers E. Functional strength measurement in cerebral palsy: feasibility, test-retest reliability, and construct validity. Dev Neurorehabil. 2019 Oct;22(7):453-461. doi: 10.1080/17518423.2018.1518963. Epub 2018 Sep 12. PMID 30207812
- [Background] Cappellini G, Sylos-Labini F, Assenza C, Libernini L, Morelli D, Lacquaniti F, Ivanenko Y. Clinical Relevance of State-of-the-Art Analysis of Surface Electromyography in Cerebral Palsy. Front Neurol. 2020 Dec 11;11:583296. doi: 10.3389/fneur.2020.583296. eCollection 2020. PMID 33362693